CLINICAL TRIAL: NCT04769180
Title: Extraintestinal Manifestations in Non Celiac Wheat Sensitivity
Brief Title: Extraintestinal Non Celiac Wheat Sensitivity
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, Principal Investigator, University of Palermo
Other Study IDs: ACPM27
Record Dates: First submitted 2021-02-20; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Non-celiac Gluten Sensitivity
Keywords: Non-celiac Gluten Sensitivity; Celiac Disease; Irritable Bowel Syndrome
MeSH Terms: conditions — Celiac Disease; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients affected with NCWS: 100 patients with a definitive diagnosis of NCWS, based on DBPC gluten/wheat challenge.
  Interventions: Other: Evaluation of extraintestinal manifestations
- Patients affected with CD: 50 patients affected with CD, sex- (± 5%) and age-matched (± 2 years) with the NCWS patients, selected at random during the study period.
  Interventions: Other: Evaluation of extraintestinal manifestations
- Patients affected with IBS not related to NCWS or other food allergies/intolerances: 50 patients affected with IBS, according to the Rome IV criteria, not related to NCWS or other food allergies/intolerances, sex- (± 5%) and age-matched (± 2 years) with the NCWS patients, selected at random during the study period.
  Interventions: Other: Evaluation of extraintestinal manifestations

INTERVENTIONS:
Other: Evaluation of extraintestinal manifestations — The researchers evaluated the prevalence and kind of extraintestinal symptoms in NCWS patients and the possible relationship between the clinical, serological, genetic and histological characteristics of the NCWS patients and the number and kind of extraintestinal manifestations, using, as control groups, CD and IBS patients.
  Other Names: Extraintestinal manifestations

SUMMARY:
Non Celiac Gluten Sensitivity (NCGS), or, better, Non Celiac Wheat Sensitivity (NCWS), since it is not known the real pathogenetic component(s) of grain, is a syndrome characterized by a cohort of symptoms, both gastrointestinal and extraintestinal, related to the ingestion of gluten/wheat-containing food in subjects who are not affected by celiac disease (CD) or wheat allergy. In particular, the possibility of extraintestinal manifestations in this condition has been suggested by some reports. In most cases, they are characterized by vague symptoms, such as headache, 'foggy mind', fatigue, joint and muscle pain, leg or arm numbness (i.e., fibromyalgia-like symptoms), even if more specific complaints have been described. A possible neurological involvement has been underlined by NCWS association with gluten encephalopathy, gluten ataxia, and gluten peripheric neuropathy. NCWS patients may show even psychiatric diseases, such as anxiety, depression, and psychosis. Other described extraintestinal manifestations are dermatitis, (eczema or skin rash), gynecological disorders, and anemia. In addition, the association of NCWS with autoimmune diseases, such as autoimmune thyroiditis, and presence of anti-nuclear or other autoantibodies has been demonstrated, suggesting that, similarly to CD, NCWS might be considered as an immune system-related disease, and this aspect should be of relevance. In conclusion, the novelty of this matter has generated an expansion of literature data about the clinical features of the disease, with the unavoidable consequence that some reports are often based on low levels of evidence. The aims of the present study were to: a) retrospectively evaluate the prevalence and kind of extraintestinal symptoms in a large cohort of NCWS patients; b) to research for a possible relationship between the clinical, serological, genetic and histological characteristics of the NCWS patients and the number and kind of extraintestinal manifestations. As control groups, the researchers used CD and Irritable Bowel Syndrome (IBS) patients unrelated to NCWS or other food allergies/intolerances.

DETAILED DESCRIPTION:
Non Celiac Gluten Sensitivity (NCGS), or, better, Non Celiac Wheat Sensitivity (NCWS), since it is not known the real pathogenetic component(s) of grain, is a syndrome characterized by a cohort of symptoms, both gastrointestinal and extraintestinal, related to the ingestion of gluten/wheat-containing food in subjects who are not affected by celiac disease (CD) or wheat allergy. In detail, NCWS is distinguished by symptoms that typically take place soon after gluten/wheat ingestion, withdraw with gluten/wheat exclusion, and relapse following gluten/wheat challenge (i.e., double-blinded placebo-controlled, DBPC, gluten/wheat challenge, used for diagnostic purpose) within hours or days. The gastrointestinal clinical picture of NCWS is a combination of irritable bowel syndrome (IBS)-like manifestations, such as abdominal pain, bloating, diarrhea, or constipation, or alternation of diarrhea and constipation, and dyspepsia like-symptoms, such as postprandial heaviness, early satiety, and epigastric pain or burning. However, the possibility of extraintestinal manifestations in this condition has been suggested by some reports. In most cases, they are characterized by vague symptoms, such as headache, 'foggy mind', fatigue, joint and muscle pain, leg or arm numbness (i.e., fibromyalgia-like symptoms), even if more specific complaints have been described. A possible neurological involvement has been underlined by NCWS association with gluten encephalopathy, gluten ataxia, and gluten peripheric neuropathy. NCWS patients may show even psychiatric diseases, such as anxiety, depression, and psychosis. Other described extraintestinal manifestations are dermatitis, (eczema or skin rash), gynecological disorders, and anemia. In addition, the association of NCWS with autoimmune diseases, such as autoimmune thyroiditis, and presence of anti-nuclear or other autoantibodies has been demonstrated, suggesting that, similarly to CD, NCWS might be considered as an immune system-related disease, and this aspect should be of relevance. In conclusion, the novelty of this matter has generated an expansion of literature data about the clinical features of the disease, with the unavoidable consequence that some reports are often based on low levels of evidence. Therefore, only studies performed on large samples, with the inclusion of control groups, may be able to clearly establish whether the large information from the literature regarding extraintestinal NCWS manifestations could be supported by evidence-based agreements. Therefore, the aims of the present study were to: a) retrospectively evaluate the prevalence and kind of extraintestinal symptoms in a large cohort of NCWS patients, diagnosed by DBPC gluten/wheat challenge; b) to research for a possible relationship between the clinical, serological, genetic and histological characteristics of the NCWS patients and the number and kind of extraintestinal manifestations. As control groups, the researchers used CD and IBS patients unrelated to NCWS or other food allergies/intolerances.

ELIGIBILITY:
NCWS Inclusion Criteria:

NCWS was diagnosed after CD or WA had been ruled out in all the studied patients according to the following criteria:

* (1) negative serum assays for serum CD-anti-tissue transglutaminase (anti-tTG) immunoglobulin (Ig) A and anti-deamidated gliadin peptide (anti-DGP) IgG antibodies; (2) absence of intestinal villous atrophy, documented in all the patients carrying the DQ2 and/or the DQ8 HLA haplotypes (thus irrespective of CD-specific serum antibody negativity), evaluated when patients had a minimum intake of 100 g of wheat daily since at least 2 weeks; (3) negative IgE-mediated immune-allergy tests to wheat (skin prick tests and/or specific serum IgE detection); (4) resolution of symptoms on a standard elimination diet, without wheat, cow's milk, yeast, and other food(s) causing self-reported symptoms, followed by symptom reappearance on a DBPC wheat challenge. Additional inclusion criteria were: age older than 18 years, follow-up duration longer than 12 months after the initial diagnosis, and at least 2 outpatient visits during the follow-up period.

NCWS Exclusion Criteria:

* (1) positive anti-endomysial antibodies (EmA) in the culture medium of the duodenal biopsies, also in the case of normal villi/crypts ratio in the duodenal mucosa; (2) self-exclusion of wheat from the diet and refusal to reintroduce it before entering the study; (3) other previously diagnosed gastrointestinal disorders; (4) nervous system disease and/or major psychiatric disorder; (5) physical impairment limiting physical activity.

CD Inclusion Criteria:

* (1) positive serum anti-tTG and EmA IgA and IgG antibodies; (2) presence of intestinal villous atrophy.

CD Exclusion Criteria:

* (1) self-exclusion of wheat from the diet and refusal to reintroduce it before entering the study; (2) other previously diagnosed gastrointestinal disorders; (3) nervous system disease and/or major psychiatric disorder; (4) physical impairment limiting physical activity.

IBS Inclusion Criteria:

* IBS diagnosis was made in accordance with the Rome IV criteria. None of these patients improved on the same standard elimination diet followed by the patients with NCWS for 4 weeks, thus confirming that the IBS diagnosis was unrelated to NCWS or other food allergies/intolerances. The patients kept a food diary during the elimination diet period to monitor their adherence to the diet; patients who did not strictly adhere to the elimination diet were not included in this study group. In patients with a diarrhea-predominant IBS presentation, the exclusion of other diagnoses was based on the assays recently suggested by the American Gastroenterology Association

IBS Exclusion Criteria:

* (1) self-exclusion of wheat from the diet and refusal to reintroduce it before entering the study; (2) other previously diagnosed gastrointestinal disorders; (3) nervous system disease and/or major psychiatric disorder; (4) physical impairment limiting physical activity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The researchers evaluated the extraintestinal manifestations in 3 groups of patients: (1) 100 patients with a definitive diagnosis of NCWS, based on DBPC gluten/wheat challenge; (2) 50 patients affected with CD, sex- (± 5%) and age-matched (± 2 years) with the NCWS patients, selected at random during the study period; (3) 50 patients affected with IBS, according to the Rome IV criteria, not related to NCWS or other food allergies/intolerances, sex- (± 5%) and age-matched (± 2 years) with the NCWS patients, selected at random during the study period.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of extraintestinal symptoms in NCWS patients | Up to 15 years
  Evaluation of systemic (malaise, fatigue), dermatological (eczema or skin rash), neurological (headache, 'foggy mind', gluten encephalopathy, gluten ataxia, gluten peripheric neuropathy, leg or arm numbness), psychiatric (anxiety, depression, psychosis), musculoskeletal (joint and muscle pain), gynaecological, and hematological (anemia) symptoms in NCWS patients.
Evaluation of extraintestinal symptoms in CD patients | Up to 15 years
  Evaluation of systemic (malaise, fatigue), dermatological (eczema or skin rash), neurological (headache, 'foggy mind', gluten encephalopathy, gluten ataxia, gluten peripheric neuropathy, leg or arm numbness), psychiatric (anxiety, depression, psychosis), musculoskeletal (joint and muscle pain), gynaecological, and hematological (anemia) symptoms in CD patients.
Evaluation of extraintestinal symptoms in IBS patients unrelated to NCWS or other food allergies/intolerances. | Up to 15 years
  Evaluation of systemic (malaise, fatigue), dermatological (eczema or skin rash), neurological (headache, 'foggy mind', gluten encephalopathy, gluten ataxia, gluten peripheric neuropathy, leg or arm numbness), psychiatric (anxiety, depression, psychosis), musculoskeletal (joint and muscle pain), gynaecological, and hematological (anemia) symptoms in IBS patients unrelated to NCWS or other food allergies/intolerances.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, MD, Principal Investigator — University of Palermo
Locations (2):
- Italy (2):
  - Internal Medicine Division of the "Cervello-Villa Sofia" Hospital, Palermo, PA
  - Department of Internal Medicine, University Hospital of Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mansueto P, Soresi M, Candore G, Garlisi C, Fayer F, Gambino CM, La Blasca F, Seidita A, D'Alcamo A, Lo Sasso B, Florena AM, Geraci G, Caio G, Volta U, De Giorgio R, Ciaccio M, Carroccio A. Autoimmunity Features in Patients With Non-Celiac Wheat Sensitivity. Am J Gastroenterol. 2021 May 1;116(5):1015-1023. doi: 10.14309/ajg.0000000000000919. PMID 33009065
- [Result] Soresi M, Incandela S, Mansueto P, Incandela G, La Blasca F, Fayer F, D'Alcamo A, Florena AM, Carroccio A. Gynecological Disorders in Patients with Non-celiac Wheat Sensitivity. Dig Dis Sci. 2021 Jan;66(1):167-174. doi: 10.1007/s10620-020-06184-8. Epub 2020 Mar 7. PMID 32146601
- [Result] Mansueto P, Soresi M, La Blasca F, Fayer F, D'Alcamo A, Carroccio A. Body Mass Index and Associated Clinical Variables in Patients with Non-Celiac Wheat Sensitivity. Nutrients. 2019 May 29;11(6):1220. doi: 10.3390/nu11061220. PMID 31146428
- [Result] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Result] Carroccio A, Giambalvo O, Blasca F, Iacobucci R, D'Alcamo A, Mansueto P. Self-Reported Non-Celiac Wheat Sensitivity in High School Students: Demographic and Clinical Characteristics. Nutrients. 2017 Jul 19;9(7):771. doi: 10.3390/nu9070771. PMID 28753927
- [Result] Carroccio A, Soresi M, D'Alcamo A, Sciume C, Iacono G, Geraci G, Brusca I, Seidita A, Adragna F, Carta M, Mansueto P. Risk of low bone mineral density and low body mass index in patients with non-celiac wheat-sensitivity: a prospective observation study. BMC Med. 2014 Nov 28;12:230. doi: 10.1186/s12916-014-0230-2. PMID 25430806
- [Result] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240